CLINICAL TRIAL: NCT06856291
Title: Treatment Response to Incretin Mimetics in Non-diabetic Obese Patients With and Without Insulin Resistance (TRIM-IR)
Brief Title: Response to Semaglutide in Non-diabetic Obese Patients With Varying Degrees of Insulin Resistance
Acronym: TRIM-IR
Status: Recruiting | Type: Observational
Sponsor: ETH Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-02395
Record Dates: First submitted 2025-02-18; First posted 2025-03-04 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: Obesity and Obesity-related Medical Conditions; Obesity and Overweight; Insulin Sensitivity/Resistance; Semaglutide
Keywords: Insulin Resistance; incretin mimetics; semaglutide; weight loss; adipose tissue function; obesity; hyperinsulinemic euglycemic clamp; obesity management; insulin sensitivity
MeSH Terms: conditions — Obesity; Overweight; Insulin Resistance; Weight Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood analyses (EDTA, Hep, glucose measurement throughout clamp test) Adipose tissue biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Non-diabetic obese individuals on semaglutide for weight loss: Non-diabetic obese individuals with planned semaglutide treatment as a weight loss intervention

SUMMARY:
Incretin mimetics are widely used pharmacological treatments for weight loss, known for their high efficacy and favorable safety profile. As the most commonly prescribed drug in this class, semaglutide is effective in both diabetic and non-diabetic individuals. However, treatment responses vary significantly, with non-diabetic individuals typically experiencing better weight loss outcomes. Despite this, up to 10% of non-diabetic individuals show little or no response to treatment, and the reasons for this variability remain unclear.

The TRIM-IR study aims to investigate the role of insulin resistance (IR) in weight loss outcomes among non-diabetic obese individuals receiving semaglutide. This single-center, observational study will assess the impact of IR on weight loss, body composition, and adipose tissue function during the first 16 weeks of semaglutide therapy. The study will also explore molecular markers of adipose tissue dysfunction, focusing on the transition from dysfunctional to healthy adipose tissue.

The investigators hypothesize, that individuals with lower IR will experience greater weight loss than those with higher IR, and that the glucose infusion rate (GIR) during hyperinsulinemic euglycemic clamp testing will correlate with weight loss variability. Secondary objectives include comparing changes in fat and lean mass, reductions in visceral fat, and improvements in adipose tissue function before and after 16 weeks of treatment. Exploratory analyses will assess adipocyte subpopulations and their response to insulin sensitivity changes.

A total of 40 participants, equally distributed by gender, will be enrolled to ensure statistical power for detecting clinically relevant differences. The study aims to optimize semaglutide use for personalized obesity treatment and provide insights into the relationship between obesity, insulin resistance, and adipose tissue plasticity, with implications for improving obesity management and cardiovascular health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60 years
2. BMI 30 - 40 kg/m2

   a. Participants must meet the eligibility criteria for coverage under the KVG (Federal Health Insurance Act) and the Specialties List, which include a weight-related comorbidity (arterial hypertension, dyslipidemia) for participants with a BMI of 30- 35 kg/m2
3. Planned therapy with semaglutide as a weight loss intervention
4. No known presence of a diabetic state
5. Ability to understand and sign a Patient Information and Consent Form

Exclusion Criteria:

1. Pregnancy or active breast feeding

   1. Therapy with semaglutide is not approved for use during pregnancy or while breastfeeding, as its safety and efficacy in these conditions have not been established.
   2. Pregnancy is an exclusion criterion for the planned investigations to avoid placing pregnant individuals under unnecessary physical or psychological stress that could pose risks to both the individual and the fetus.
2. Medication and/or pathologies that prevent the safe execution of the fat tissue biopsies (e.g. allergy towards local anesthetics, disorders of coagulation, treatment with anticoagulants)
3. Medical conditions that prevent examinations and testing (e.g. epilepsia, symptomatic cardiovascular disease)
4. History of or planned bariatric surgery
5. HbA1c ≥ 6.5% as measured by the central laboratory at screening
6. Fasting plasma-glucose >7.0 mmol/l
7. History of type 1 or type 2 diabetes mellitus
8. Treatment with glucose-lowering agent(s) (e.g. Metformin) within 90 days before screening
9. Treatment with a GLP-1 (glucagon like peptide 1) receptor agonist within 180 days before screening
10. A self-reported change in body weight >5% within 90 days before screening
11. Active malignancy (<2a since remission)
12. Treatment with any medication for the indication of obesity within the past 90 days before screening
13. Uncontrolled thyroid disease, defined as thyroid stimulating hormone (TSH) > 10 mIU/L or < 0.4 mIU/L as measured by the central laboratory at screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Planned gender distribution of females:males is 1:1, determined by biological sex
Study Population: The investigators plan to include a total of 40 non-diabetic, obese individuals that will undergo treatment with semaglutide as a weight-loss intervention independent of our observational study. To avoid a highly heterogeneous participant group, inclusion in the study will be limited to individuals with a BMI between 30 and 40 kg/m². Patients with a prediabetic state will not be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in body weight (%) | 16 weeks

SECONDARY OUTCOMES:
Change in fat mass (%) | 16 weeks
  measured by DEXA (dual energy x-ray absorptiometry)
Change in lean mass (%) | 16 weeks
  measured by DEXA
Change in abdominal visceral fat area (in cm2) | 16 weeks
  measured by DEXA

OTHER OUTCOMES:
Change in cell size of adipose tissue after 16 weeks of semaglutide treatment | 16 weeks
  The size of adipocytes is a direct measure of adipose tissue quality and function. It will be evaluated through histological examinations.
Changes in cell distribution of adipose tissue after 16 weeks of semaglutide treatment | 16 weeks
  Changes in the distribution of adipocytes and other components of adipose tissue (e.g. macrophages, progenitors) serve as a direct measure of adipose tissue quality and function. It will be evaluated through histological examinations.
Changes in signs of fibrosis in adipose tissue after 16 weeks of semaglutide treatment | 16 weeks
  Signs of fibrosis are a direct measure of adipose tissue quality and function. They will be evaluated through histopathological analysis.
Changes in inflammatory activity of adipose tissue after 16 weeks of semaglutide treatment | 16 weeks
  Inflammatory activity, measured by the number and type of white blood cells infiltrating adipose tissue, is a direct way to assess adipose tissue quality and function. It will be evaluated by quantifying inflammatory cells within the tissue.
Change in adipokine secretion pattern after 16 weeks of semaglutide treatment | 16 weeks
  The adipokine-secretion pattern is an indirect way to assess adipose tissue quality and function. We will analyze leptin, adipokines, and other relevant markers in blood samples and potentially in adipose tissue from strong or weak responders to identify patterns that may help predict significant changes or the absence of response.
Change in systemic inflammation after 16 weeks of semaglutide treatment | 16 weeks
  Adipose tissue dysfunction can contribute to systemic inflammation, making it an indirect measure of adipose tissue quality. Serum levels of systemic inflammatory markers such as C-reactive protein (CRP), interleukins, and tumor necrosis factor-alpha (TNF-α) will be assessed before and after 16 weeks of semaglutide treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Wolfrum, Prof. Dr., Study Chair — ETH Zurich
Locations (1):
- Cantonal Hospital Aarau, Aarau, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided